CLINICAL TRIAL: NCT05470413
Title: A Randomized, Double-Blinded, and Placebo-Controlled Phase III Study to Evaluate the Efficacy and Safety of SHR0302 in Adult Patients With Severe Alopecia Areata
Brief Title: Evaluate the Efficacy and Safety of SHR0302 in Adult Patients With Severe Alopecia Areata
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Reistone Biopharma Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RSJ10535
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata | interventions — ivarmacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHR0302 4 mg (Active Comparator): Drug：SHR0302
  Interventions: Drug: SHR0302
- SHR0302 8 mg (Active Comparator): Drug：SHR0302
  Interventions: Drug: SHR0302
- Placebo (Placebo Comparator): Drug: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHR0302 — SHR0302 4 mg
  Arms: SHR0302 4 mg
Drug: SHR0302 — SHR0302 8 mg
  Arms: SHR0302 8 mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a multi-central, double-blind, randomized, parallel, placebo-controlled phase 3 study in adult subjects with severe alopecia areata (SALT≥50%). Approximately 330 adult patients will be enrolled into the study. Efficacy and safety of two doses of SHR0302 will be compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects with the age of ≥18 and ≤ 65 years old at the time of informed consent
2. Have severe alopecia areata (AA), as determined by all of the followings:

   1. Clinical diagnosis of AA with no other cause of hair loss;
   2. ≥ 50% scalp involvement of alopecia (using SALT score), including alopecia totalis (AT) and alopecia universalis (AU). AT refers to scalp hair loss SALT 95-100 (both inclusive) and AU refers to scalp hair loss SALT 95-100 (both inclusive), plus facial or body hair loss.
   3. Duration of the current episode of scalp hair loss of at least 6 months and less than 8 years, and without terminal hair regrowth within 6 months prior to screening and baseline
3. All women of childbearing potential and all men must be willing to use at least one highly effective method of contraception from the signing of informed consent, throughout the duration of the study, and for 4 weeks after the last dose of investigational drugs.
4. Capable of providing a signed and dated informed consent form indicating the subject has been fully informed, and are willing to comply with the scheduled visits, treatment plan, laboratory testing, and other study procedures.

Exclusion Criteria:

1. Alopecia caused by other reasons, including but not limited to syphilitic alopecia, androgenetic alopecia (AGA), scarring alopecia, diffuse alopecia (manifested as diffuse hair loss), serpiginous alopecia areata (involving the temporal and occipital hairline), traction alopecia, anagen effluvium, folliculotropic mycosis fungoides (FMF), or hair loss caused by thyroid diseases.
2. Any other active skin disease, scalp disorder, or active scalp trauma, that in the opinion of the investigator would interfere with study assessments of efficacy or safety. Subjects with shaved heads must not enter the study until the hair has grown back and is considered stable by the investigator.
3. Have received any of the following treatment within the specified timeframes:

   •Previously systemic treated with JAK inhibitors, e.g., tofacitinib, baricitinib, upadacitinib, PF04965842, and ritlecitinib (PF-06651600).

   Exception: Patients with previous use of topical JAK inhibitors for diseases other than AA (non-scalp sites) were allowed. (discontinued 8 weeks prior to the first dose).
   * Any of the below treatments within 8 weeks prior to the first dose of investigational drugs: topical immunotherapy, e.g., diphenylcyclopropenone (DPCP); systemic treatment to AA, e.g., oral or intravenous corticosteroids, cyclosporin; and intralesional immunosuppressant therapy.
   * Any of the below treatments within 4 weeks or 5 half-lives of the drug (if known) prior to the first dose of investigational drugs, whichever is longer: topical treatments, phototherapy, cryotherapy, or any other treatment to AA.
4. Subjects have potential active, latent, or inadequately treated infection of tubercle bacillus (TB, including, but not limited to pulmonary TB), as evidenced by any of the followings:

   * Subjects is currently being treated for active TB infection.
   * Positive QuantiFERON-TB Gold (QFT Gold test) or T-SPOT test or other interferon-gamma release assays (IGRAs) test performed within 3 months prior to/within the screening period, and those who have negative results of above tests but with clinical symptoms and/or abnormal chest X-ray that could not exclude TB infection;
   * History of either untreated or inadequately treated latent or active TB infection.

   Exception: Subject with a history of active TB who has documented evidence of appropriate treatment, has no history of re-exposure since his/her treatment was completed, and has a screening chest x-ray with no evidence of active TB may be enrolled if other entry criteria are met. Such subject would not be required to undergo the protocolspecific TB testing for QuantiFERON®-TB Gold test, or T-SPOT.TB test or other interferon-gamma release assays (IGRAs) test but must have a chest x-ray at screening.
5. Subjects who currently have thyroid disorders (abnormal TSH levels at screening with associated abnormal fT4 or fT3 values, including hyperthyroidism and hypothyroidism), in the opinion of the investigator, pose an unacceptable risk for the patient's participation in the study.

   Note: Patients who are receiving thyroxine as replacement therapy may participate in the study, provided stable therapy has been administered for

   ≥12 weeks and TSH is within the laboratory's reference range. Patients who are receiving stable thyroxine replacement therapy who have TSH marginally outside the laboratory's normal reference range may participate if the treating physician has documented that the thyroxine replacement therapy is adequate for the patient.
6. Subjects with a history of thrombotic disease.
7. Subjects who may receive immunization with any live or attenuated vaccine within 4 weeks before the first dose of investigational drugs.
8. Subjects who have participated in clinical trials of any drug or medical device within the last 1 month or 5 half-lives of the drug (whichever is longer) before screening
9. Subjects with a history of severe neuropsychiatric disorders.
10. Subjects with evidence of clinical laboratory abnormalities at screening that, in the opinion of the investigator, may affect the safety of subjects or the interpretation of study results:

    1. Hemoglobin level < 9.0 g/dL or hematocrit < 30%.
    2. Absolute white blood cell (WBC) count < 3.0 × 109/L (< 3000/mm3) or absolute neutrophil count (ANC) < 1.2 × 109/L (< 1200/mm3).
    3. Thrombocytopenia, as defined by a platelet count of < 100 × 109/L (< 100,000/mm3).
    4. Total bilirubin, alkaline phosphatase (ALP), aspartate aminotransferase (AST), or alanine aminotransferase (ALT) > 2 × ULN. subjects with hepatic cirrhosis will be excluded.
    5. Subjects with eGFR ≤ 60 mL/min based on Cockcroft-Gault calculation, or patients currently undergoing regular hemodialysis or peritoneal dialysis.
11. Screening 12-lead ECG that demonstrates clinically relevant abnormalities which, in the opinion of the investigator, may affect subject safety or would interfere with study assessments if being enrolled into the study.
12. Subject with the following concurrent or previous conditions:

    1. Clinically significant infections (e.g., requiring hospitalization or parenteral antibiotics) or opportunistic infections within 1 month prior to baseline,
    2. History of more than one episode of herpes zoster or disseminated herpes zoster (single episode) infection,
    3. Any other infections that, in the opinion of the investigator, may aggravate if the subject participate in the study,
    4. Any infection requiring antibacterial treatments within 2 weeks of randomized.
13. Women who are pregnant or lactating or planning pregnancy while enrolled in the study. Male subjects who are planning to donate sperm during the study or within 4 weeks after the last dose of investigational drugs.
14. History of alcohol or drug abuse with less than 6 months of abstinence prior to baseline, and unsuitable for the study in the opinion of the investigator.
15. Subjects with a history of hypersensitivity or allergies to JAKi, any of its ingredients, or similar compounds.
16. Subjects with malignancies/lymphadenosis or a history of malignancies/lymphadenosis, except for adequately treated or excised non-metastatic basal cell or squamous cell carcinoma of the skin.
17. Subjects with positive specific treponema pallidum antibody, human immunodeficiency virus (HIV), or hepatitis B/C virus:

    1. HBV positive: HBsAg positive or HBcAb positive + HBV DNA positive. NOTE: Subjects with HBcAb positive + HBV DNA negative can participate in the study.
    2. HCV positive: HCV antibody positive + HCV RNA positive. NOTE: Subjects with HCV antibody positive+ HCV RNA negative can participate in the study.
    3. HIV positive: HIV antibody positive.
18. Any other condition which in the opinion of the investigator would make the subject unsuitable for inclusion in the study.
19. With evidence of clinically significant cardiovascular, mental, renal, hepatic, immune, gastrointestinal, urogenital, nervous system, musculoskeletal, cutaneous, sensory, endocrine (including uncontrolled diabetes or thyroid disease), or hematologic abnormalities. A clinically significant disease is defined as any disease that in the opinion of the investigator will endanger the safety of a subject during the participation, or the disease/condition may worsen during the study and affect the efficacy or safety analysis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-02-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects achieving a SALT score ≤ 20 at week 24 | 24 weeks
  Percentage of subjects achieving a SALT score ≤ 20 at week 24

SECONDARY OUTCOMES:
Percentage of subjects achieving a 50% improvement in SALT score (SALT50) at Week 24. | 24 weeks
  Percentage of subjects achieving a 50% improvement in SALT score (SALT50) at Week 24.
Percentage of subjects with a SALT score ≤ 20 at Weeks 4, 8, 12, 16, 28, 36, 44, and 52. | Weeks 4, 8, 12, 16, 28, 36, 44, and 52
  Percentage of subjects with a SALT score ≤ 20 at Weeks 4, 8, 12, 16, 28, 36, 44, and 52.
Percentage of subjects achieving a 50% improvement in SALT score (SALT50) at Weeks 4, 8, 12, 16, 28, 36, 44, and 52. | Weeks 4, 8, 12, 16, 28, 36, 44, and 52.
  Percentage of subjects achieving a 50% improvement in SALT score (SALT50) at Weeks 4, 8, 12, 16, 28, 36, 44, and 52.
Percentage of subjects achieving a 75% improvement in SALT score (SALT75) at Weeks 4, 8, 12, 16, 24, 28, 36, 44, and 52. | Weeks 4, 8, 12, 16, 24, 28, 36, 44, and 52.
  Percentage of subjects achieving a 75% improvement in SALT score (SALT75) at Weeks 4, 8, 12, 16, 24, 28, 36, 44, and 52.
Percentage of subjects achieving a 90% improvement in SALT score (SALT90) at Weeks 4, 8, 12, 16, 24, 28, 36, 44, and 52. | Weeks 4, 8, 12, 16, 24, 28, 36, 44, and 52.
  Percentage of subjects achieving a 90% improvement in SALT score (SALT90) at Weeks 4, 8, 12, 16, 24, 28, 36, 44, and 52.
Absolute change from baseline in SALT score at Weeks 4, 8, 12, 16, 24, 28, 36, 44, and 52. | Weeks 4, 8, 12, 16, 24, 28, 36, 44, and 52.
  Absolute change from baseline in SALT score at Weeks 4, 8, 12, 16, 24, 28, 36, 44, and 52.
Percentage change from baseline in SALT score at Weeks 4, 8, 12, 16, 24, 28, 36, 44, and 52. | Weeks 4, 8, 12, 16, 24, 28, 36, 44, and 52.
  Percentage change from baseline in SALT score at Weeks 4, 8, 12, 16, 24, 28, 36, 44, and 52.
Percentage of subjects with an absolute SALT score ≤ 10 at Weeks 4, 8, 12, 16, 24, 28, 36, 44, and 52. | Weeks 4, 8, 12, 16, 24, 28, 36, 44, and 52.
  Percentage of subjects with an absolute SALT score ≤ 10 at Weeks 4, 8, 12, 16, 24, 28, 36, 44, and 52.
Percentage of subjects achieving "Satisfied" in Subject's Global Assessment (SGA) at Weeks 24, 36, and 52. | Weeks 24, 36, and 52.
  Percentage of subjects achieving "Satisfied" in Subject's Global Assessment (SGA) at Weeks 24, 36, and 52.

CONTACTS AND LOCATIONS:
Locations (31):
- China (31):
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Chongqing Traditional Chinese Medicine Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guanzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Wuhan No.1 Hospital, Wuhan, Hubei
  - The second xiangya hospital of central south university, Changsha, Hunan
  - Xiangya Hospital Of Central South University, Changsha, Hunan
  - Dermatology Hospital of Chinese Academy of Medical Sciences, Nanjing, Jiangsu
  - Jiangsu Province People's Hospital, Nanjing, Jiangsu
  - Wuxi No.2 People's Hospital, Wuxi, Jiangsu
  - Jiangxi Provincial Hospital of Dermatology, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital Of China Medical University, Shengyang, Liaoning
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality
  - First Hospital Of Shanxi Medical University, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Hangzhou Third People's Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital Of Zhejiang Chinese Medical University, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang